CLINICAL TRIAL: NCT06622356
Title: Multivariate Analysis and Machine Learning Model Risk Prediction of Recurrent Pain After PLIF Surgery for Degenerative Lumbar Spine Disease At Long-term Follow-up
Status: Completed | Type: Observational
Sponsor: Hao Liu (Other)
Responsible Party: Sponsor-Investigator, Hao Liu, Orthopedic surgeon, First Affiliated Hospital of Suzhou University, Jiangsu Province, China, First Affiliated Hospital of Suzhou Medical College
Organization: First Affiliated Hospital of Suzhou Medical College (Other)
Other Study IDs: (2024) Lun Yan Grant No. 517; (2024) Lun Yan Grant No. 517 (Other: Medical Ethics Committee of the First Affiliated Hospital of Soochow University)
Record Dates: First submitted 2024-09-28; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Lumbar Disc Herniation; Lumbar Degenerative Disease; Sarcopenia
Keywords: Lumbar Degenerative disease; PLIF; Sarcopenia; Sagittal balance; Machine learning; SVM; Cross Validation
MeSH Terms: conditions — Intervertebral Disc Displacement; Sarcopenia | interventions — Magnetic Resonance Spectroscopy; gadolinium ethoxybenzyl DTPA

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Biological samples were not designed for this study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Rehabilitation Group: Rehabilitation Group (n = 268): mild/non pain group with VAS<3 at 12-18 months after PLIF。The study was retrospective and did not design an intervention
  Interventions: Other: MRI with Eovist
- Recurrent pain group: Recurrent pain group (n = 184): recurrent pain group with VAS≥3 at 12-18 months after PLIF
  Interventions: Other: MRI with Eovist

INTERVENTIONS:
Other: MRI with Eovist — The study was retrospective and did not design an intervention

SUMMARY:
The study was a clinical retrospective study designed to investigate risk factors for long-term recurrent pain after PLIF in patients with lumbar degenerative disease and to improve patient outcomes

ELIGIBILITY:
Inclusion Criteria:

1. confirmed diagnosis of lumbar degenerative disease (spinal stenosis, disc herniation with lumbar instability, and lumbar spondylolisthesis), with no significant symptomatic relief after conservative treatment for more than 3 months, and in need of surgical intervention;
2. lumbar spinal fusion surgical treatment with PLIF;
3. grouping based on the presence or absence of a lumbar or limb pain with VAS ≥3 at the 12-18 month postoperative follow-up;
4. observational indicators including individual factors, surgical factors, spine-pelvis sagittal balance parameters, and paravertebral muscle parameters.

Exclusion Criteria:

(1) those with a history of lumbar spine trauma, inflammation, tumor, or surgery; (2) those with congenital or acquired severe lumbar vertebral deformity; (3) those with severe neurological dysfunction; (4) those with incomplete baseline and follow-up data.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study retrospectively reviewed 452 patients suffering from degenerative lumbar spinedisorders in our institute between January 2019 and February 2023. The patients were separated into Recurrent pain group and Rehabilitation Group. Recurrent pain group (n = 268): mild/non pain group with VAS<3 at 12-18 months after PLIF；Rehabilitation Group (n = 184): recurrent pain group with VAS≥3 at 12-18 months after PLIF.
Sampling Method: Non-Probability Sample
Enrollment: 452 (Actual)
Dates: Start 2024-09-20 (Actual); Primary Completion 2024-09-25 (Actual); Study Completion 2024-09-28 (Actual)

PRIMARY OUTCOMES:
SAS（Pain rating scale） | 12-18 months after surgery
  The visual analogue scale (VAS) was employed to determine the patient's perception of lower back pain or lower limb pain prior to surgery, as well as 12-18 months after surgery. (0-10 scale, with 0 being painless and 10 being the most painful)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical record system and imaging system of the First Affiliated Hospital of Suzhou University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
Before January 1,2025;in the form of paper.The original data of the trial will be uploaded to Genome Sequence Archive (GSA) (ngdc.cncb.ac.cn)